CLINICAL TRIAL: NCT01908764
Title: An Open-Label, Single Dose, Pharmacokinetic Study of AL-60371 Otic Suspension, 0.3% in Pediatric Subjects Following Tympanostomy Tube Surgery
Brief Title: Pharmacokinetic Study of AL-60371 Otic Suspension in Pediatric Subjects Following Tympanostomy Tube Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C-13-023
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2014-10

CONDITIONS: Otitis Media
Keywords: ear tubes; tympanostomy tubes; Otitis Media at the time of Tympanostomy Tube surgery; OMTT
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-60371/Posology 1 (Experimental): AL-60371 otic suspension, single dose of 200 µL following surgical insertion of tympanostomy tubes
  Interventions: Drug: AL-60371 otic suspension
- AL-60371/Posology 2 (Experimental): AL-60371 otic suspension, single dose of 4 drops following surgical insertion of tympanostomy tubes
  Interventions: Drug: AL-60371 otic suspension

INTERVENTIONS:
Drug: AL-60371 otic suspension

SUMMARY:
The purpose of this study is to describe the pharmacokinetics of AL-60371 otic suspension following two posologies of bilateral ototopical doses in pediatric subjects immediately after bilateral tympanostomy tube surgery.

ELIGIBILITY:
Inclusion Criteria:

* Requires bilateral myringotomy and tympanostomy tube insertion;
* Provides informed consent (parent/legal guardian);
* Signs assent form where applicable (subject);
* Accompanied by parent/legal guardian at each visit;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Menarcheal females;
* Current or recent history of any disease which, in the opinion of the Principal Investigator, may place the subject at risk or interfere with study;
* Use of excluded medications within one week prior to surgery and for the duration of the study;
* Requires another surgical procedure in addition to the myringotomy;
* Clinically relevant otic condition which, in the opinion of the Principal Investigator, would preclude the safe administration of the study medication;
* Participation in any other investigational study within 30 days before entry into this study or along with this study;
* Known or suspected allergy or hypersensitivity to any active or inactive ingredient in the test article;
* Other protocol-defined exclusion criteria may apply.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Maximum observed analyte plasma concentration (Cmax) | Day 1/Surgery Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6 hours post-dose
  The analyte plasma concentrations at each collection time point will be quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS).
Time to reach Cmax (Tmax) | Day 1/Surgery Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6 hours post-dose
  The analyte plasma concentrations at each collection time point will be quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS).
Area under the analyte plasma concentration-time curve to the last quantifiable sampling time point (AUC0-last) | Day 1/Surgery Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6 hours post-dose
  The analyte plasma concentrations at each collection time point will be quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS).
Area under the concentration-time curve from 0 to infinity (AUC0-∞) | Day 1/Surgery Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6 hours post-dose
  The analyte plasma concentrations at each collection time point will be quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS).
Time to last measurable concentration (Tlast) | Day 1/Surgery Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6 hours post-dose
  The analyte plasma concentrations at each collection time point will be quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS).
The terminal elimination half (T½) | Day 1/Surgery Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6 hours post-dose
  The analyte plasma concentrations at each collection time point will be quantitated using a high performance liquid chromatography/tandem mass spectrometry method (HPLC/MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Celeste McClean, BS, MT (ASCP), Study Director — Alcon Research